CLINICAL TRIAL: NCT01115270
Title: A Study Comparing Shunt Placement Versus Endoscopic Third Ventriculostomy in the Treatment of Hydrocephalus
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Marvin Bergsneider, Marvin Bergsneider, M.D., University of California, Los Angeles
Other Study IDs: 5R01NS054881-04 (NIH); 07-08-038-03 (Other Grant/Funding Number: IRB)
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Hydrocephalus, Normal Pressure
Keywords: Normal Pressure Hydrocephalus
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hydrocephalus Patients: Those patients diagnosed with Normal Pressure Hydrocephalus.
  Interventions: Other: Non-invasive measures
- Normal Participants: Individuals who are not diagnosed with Normal Pressure Hydrocephalus.
  Interventions: Other: Non-invasive measures

INTERVENTIONS:
Other: Non-invasive measures — assessment of cerebrovascular fluid movement

SUMMARY:
The main purpose of this study is to compare two types of treatment of hydrocephalus: placement of a ventriculoperitoneal (VP) shunt versus an endoscopic third ventriculostomy (ETV). A second goal of this study will be to understand how the two different types of procedures, VP shunt versus ETV, affect brain blood flow and pressures. Understanding these changes is important because the investigators hope is to someday be able to predict who will better respond to one procedure or another.

DETAILED DESCRIPTION:
The management of normal pressure hydrocephalus (NPH) is challenging due to diagnostic uncertainties and high treatment risks. To date, there are no evidence-based treatment standards for this disorder. Our long-term goal is to improve the outcome of NPH improving our understanding of cerebrospinal fluid (CSF) hydrodynamics. The Specific Aims are to 1) determine the value of a high volume tap test, and 2) determine whether intracranial hemo/hydrodynamic variables, measured before a shunt operation, support the tuned-dynamic absorber model of intracranial pressure dynamics.

The study's Aim relates to modeling the complex hydro- and hemodynamics of intracranial physiology-pathology. We hypothesize that current hydrocephalus models are over-simplistic and that shunt-induced hydrodynamics are better modeled based on ICP waveform characteristics and the application of novel dynamic models. Much of the data for this Aim will be passively recorded during the routine care of the patient. In essence, we are only adding noninvasive MRI studies and TCD (transcranial Doppler) studies.

The experimental methodology is aimed at altering the intracranial compartment compliance by placing the patient in various positions so that these phase differences can be detected. The simplest way to alter intracranial compliance is to make postural changes. When a patient is in the Trendelenburg position, venous outflow out of the brain is hindered resulting in an increase in ICP and presumably a reduction in compliance. Conversely, raising the head of bed to 60 degrees will result in the opposite effect. The second mechanism of altering compliance (and ICP) will occur as a result of treating the hydrocephalus with a CSF shunt. Because we are able to study hydrocephalus patients prior to shunting as part of their diagnostic workup, we create a new state with the shunt that will allow us to further characterize the intracranial system.

ELIGIBILITY:
Inclusion Criteria:

* Findings of gait/balance disturbance must be present, plus at least one other area of impairment in cognition, urinary symptoms or both
* Minimum duration of symptoms of at least three months, progression over time, and no other neurological, psychiatric or general medical conditions that are sufficient to explain the presenting symptoms
* MRI or CT performed after onset of symptoms must show evidence of ventricular enlargement (Evan's index > 0.3) not entirely attributable to cerebral atrophy or congenital enlargement
* Criteria for shunt placement: we place greatest emphasis on the results of the temporary CSF drainage trial. Patients who experience a temporary improvement in neurological function (gait, bladder control, and/or cognition) are offered a shunt operation. For patients in whom the CSF drainage results were equivocal, then other factors such as elevated baseline ICP and/or high Rout will also be considered for a shunt under these circumstances

Exclusion Criteria:

* Age < 40
* Fixed musculoskeletal deformities that will exclude gait improvement
* Advanced dementia
* Inability to obtain an MRI study
* General medical conditions in which operative risks are excessive
* Patients taking Warfarin (Coumadin) will be excluded

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized NPH and non-NPH patients
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2007-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
intracranial compliance | 72 hours
  assessment of pulsatile cerbrovascular fluid movement

SECONDARY OUTCOMES:
cerebrovascular change | 72 hours
  neuroimaging

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Bergsneider, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Neurosurgery, Los Angeles, California, United States